CLINICAL TRIAL: NCT03436121
Title: Single-dose Ketamine to Reduce Pain Severity, Depressive Symptoms and the Need for Opiates Both During and After Emergency Department Care
Brief Title: Single-dose Ketamine for the Reduction of Pain and Depression in the Emergency Department
Status: Withdrawn | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: Ketamine shortage during the funding period of the trial
Sponsor: Maria Pacella (Other)
Collaborators: University of Pittsburgh Physicians (Other)
Responsible Party: Sponsor-Investigator, Maria Pacella, Assistant Professor, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PRO17090065
Record Dates: First submitted 2018-01-31; First posted 2018-02-19 (Actual); Last update posted 2020-02-11 (Actual); Status verified 2020-02

CONDITIONS: Acute Pain; Depression
MeSH Terms: conditions — Acute Pain; Depression | interventions — Ketamine; Midazolam

STUDY DESIGN:
Intervention Model Description: Participants will be randomly assigned to either the experimental condition (ketamine + midazolam) or the active control condition (placebo + midazolam)
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Experimental Arm (Experimental): Participants will be assigned to receive a single dose of IV ketamine (0.3 mg.kg) + midazolam
  Interventions: Drug: Ketamine; Drug: Midazolam
- Active Placebo Arm (Active Comparator): Participants will be assigned to receive a single dose of IV placebo + midazolam
  Interventions: Drug: Midazolam; Drug: Placebo

INTERVENTIONS:
Drug: Ketamine — Ketamine is a medication approved by the US Food and Drug Administration (FDA) for anesthesia, sedation, and post-surgical pain treatment. It is not approved for emergency patients complaining of pain but is often used "off-label." Ketamine may be useful for acute pain management and in treatment of depressed mood. The purpose of this study is to determine whether a single low dose of ketamine can relieve pain and reduce negative mood for 2 weeks after emergency department (ED) treatment.
  Arms: Experimental Arm
Drug: Midazolam — In this study, all patients will also receive midazolam. Midazolam is a sedative that typically makes people feel relaxed and is intended to increase comfort with ketamine and reduce anxiety.
Drug: Placebo — In this study, patients in the active comparator group will receive midazolam first, then placebo. A placebo is an inactive solution that looks like the study drug, but contains no active ingredients.
  Arms: Active Placebo Arm

SUMMARY:
In this proposal, the investigators will determine if a single dose of intravenous (IV) ketamine (in combination with midazolam) reduces pain severity, depressive symptoms and need for opiate analgesics both in the ED and in the acute recovery period after ED discharge. The investigators will compare the ketamine arm to an active placebo-controlled arm (with midazolam).

DETAILED DESCRIPTION:
The investigators will enroll 120 medically stable adult patients who present to two Emergency Departments with a chief complaint of acute pain.

The investigators will randomly assign subjects using a blocked randomization schedule to either: 1) a single dose of IV ketamine (0.3 mg.kg) + midazolam, or 2) placebo + midazolam. ED providers and patients will be blind to treatment allocation.

All participants will complete measures of pain and mood scores every 30 minutes, and the investigators will record any analgesics administered in the ED until discharge. At 7-days and 14-days post- discharge, the investigators will measure summary reports of pain severity, mood, and analgesic medication used.

ELIGIBILITY:
Inclusion Criteria:

1. Adults between the ages of 18-65
2. A chief complaint of painful condition (pain score ≥ 5 on the numeric rating scale [NRS] from 0-10 with anchors of 0 = "no pain" and 10 = "worst pain imaginable")
3. Expected to be in the ED for at least 2 hours

Exclusion Criteria:

1. Non-English speaking
2. Not medically suitable for ketamine per treating MD (e.g. medical condition where ketamine is contraindicated); ketamine or midazolam may be unsafe (e.g., known sensitivity, glaucoma, or other concerns)
3. Not alert and oriented
4. Active psychosis, self-injury, suicidal/homicidal intentions on initial evaluation by treating team
5. Seeking treatment due to a mental health or substance use disorder
6. History of chronic opioid use
7. Prescribed opioid use within the past 24 hours
8. Any use of recreational narcotics throughout lifetime
9. Sensitivity or allergy or intolerance to ketamine, opioids, and/or benzodiazepines
10. Weight > 170kg (375 lbs)
11. Current neurological disease (e.g., multiple sclerosis, stroke, brain tumor, seizure disorder, etc.)
12. Pregnancy
13. Prisoner

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-12 (Estimated); Primary Completion 2020-02-05 (Actual); Study Completion 2020-02-05 (Actual)

PRIMARY OUTCOMES:
Pain Intensity in the ED | Pain intensity rating in the ED at 1-hour post-study drug administration
  Pain Numeric Rating Scale (PNRS)- this item is anchored to pain intensity "right now" on a scale from 0(no pain)-10 (worst pain imaginable)

SECONDARY OUTCOMES:
Pain Intensity at Follow-Up | Pain Intensity at 1-week post-ED Discharge
  Pain Numeric Rating Scale (PNRS): this item is anchored to pain intensity within the past 7-days on a scale from 0 (no pain) to 10 (worst pain imaginable)

CONTACTS AND LOCATIONS:
Overall Officials: Maria L Pacella, PhD, Principal Investigator — University of Pittsburgh

IPD SHARING:
Plan to Share IPD: Undecided
There is no plan in place yet because it is undecided whether the investigators will need to share the data with additional investigators/researchers not listed on the protocol.